CLINICAL TRIAL: NCT02482246
Title: Coagulation Profile Surrounding Normal Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB12-1260
Record Dates: First submitted 2015-03-11; First posted 2015-06-26 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Healthy parturients presenting for scheduled cesarean delivery will have blood drawn and measured for microparticles at baseline, immediately after delivery, and at several time points thereafter.

DETAILED DESCRIPTION:
Protocol: Informed consent will be obtained and documented. Subjects who agree to participate will have an intravenous line of at least 16 gauge placed by an anesthesiologist via standard sterile technique, and lidocaine will be used for patient comfort during the procedure. The intravenous line will contain two stopcocks and will be connected to intravenous fluids as ordered by the obstetrician or anesthesiologist for patient care. If for any reason the intravenous line cannot be used for blood draws, a second intravenous line will be placed for the purpose of drawing blood samples. This line will be placed by an anesthesiologist who uses lidocaine and operates under standard sterile conditions. This line will not be connected to fluids, but to a device with a short piece of tubing used commonly for this purpose (often called a "heplock," although no heparin is used); two stopcocks will be attached to the end of this device.

Blood samples will be drawn through the intravenous line (or the "heplock" when it becomes necessary to place one) using the following procedure: a 10 mL sterile syringe will be attached to the distal stopcock and 5 mL of blood will be withdrawn (to clear the line of intravenous fluids). A second 10 mL sterile syringe will be attached to the proximal stopcock and 5 mL blood will be withdrawn for assay (total 10 mL blood withdrawn). The blood withdrawn to clear the line will be wasted. Finally, a 5 mL normal saline flush will be administered to clear the line of blood.

Blood will be drawn at baseline (placement of intravenous catheter), immediately after delivery of the placenta (within 15 minutes), 1 hour postpartum (within 1 hour and 1 hour 15 minutes), 4 hours postpartum (within 4 hours and 4 hours 15 minutes), and 24-36 hours postpartum (5 samples total per subject). After the last blood draw, the intravenous line will be discontinued if clinically indicated.

Blood will be placed in a standard "yellow top" tube and sent to the University's flow cytometry lab where it will be centrifuged and will undergo flow cytometry to measure microparticles and staining to identify endothelial-, platelet- versus leukocyte-derived microparticles and to determine placental origin. In addition Tissue Factor levels in the microparticles will be measured. Also, confirmatory image stream microscopy will be performed. Data acquisition will be performed on the ImageStreamX with validation on the Gallios Cytometer.

Demographic data collected will include age, height, weight, American Society of Anesthesiologists Physical Status Classification, gravidity, parity, estimated gestational age, and co-existing maternal or obstetric conditions. Note will be made of the date and time of each blood draw, and date and time of delivery of the baby and the placenta. Estimated blood loss will be recorded, as will blood product transfusion.

Sample size: As this is pilot data, a convenience sample of 10 patients will be studied.

Statistics: Demographic data will be presented primarily with descriptive statistics. Comparisons will be made for each assay result among the various time points (i.e., baseline values compared to values at subsequent times). Tests for normality will be performed; mean and standard deviation will be reported for normal data and median with interquartile range for non-normal data. Assay results at various time points will be compared with a mixed-model analysis of variance. A P < 0.05 will be required to reject the null hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a singleton pregnancy with gestational age greater than or equal to 36 weeks who present for scheduled cesarean delivery will be eligible for participation.

Exclusion Criteria:

* Specific exclusion criteria include emergency cesarean delivery, labor pain, hypertensive diseases of pregnancy, diabetes, known placental abnormalities such as placental abruption, placenta previa and placenta accreta, and known disorders of coagulation or recent anticoagulant therapy.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Microparticle number and type | Baseline, delivery, and 1-hr, 4-hr and 24-36-hr post delivery
  Assay of withdrawn blood

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States